CLINICAL TRIAL: NCT02817100
Title: Randomized, Placebo-controlled, Double-blind, Parallel Group Study to Investigate the Safety, Tolerability and Pharmacokinetics of Increasing Single Oral Doses (10 - 1500 mg, Tablets) of BAY1817080 Including the Effect of Food and Itraconazole on the Relative Bioavailability of BAY1817080 in Healthy Men
Brief Title: First in Human Study to Investigate the Safety and Tolerability, Pharmacokinetics, Itraconazole Drug-drug-interaction and Food Effect of BAY1817080
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 18183; 2016-000253-12 (EudraCT Number)
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Clinical Trials, Phase I as Topic
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAY1817080 (Experimental): Study Part 1: Dose 1 to 7 of BAY1817080 (increasing dose levels; redosing of BAY1817080 at dose group 1 and 2 together with itraconazole; redosing of BAY1817080 at dose group 4 together with food [American breakfast]); Study part 2: Dose 1 to 4 of BAY1817080 together with an American breakfast (increasing dose levels; redosing of BAY1817080 at dose group 1, 2 and 4 together with food [Continental breakfast])
  Interventions: Drug: BAY1817080; Drug: Itraconazole
- Placebo (Placebo Comparator): Study Part 1: Placebo Dose 1 to 7 of BAY1817080; Study Part 2: Placebo Dose 1 to 4 of BAY1817080
  Interventions: Drug: Placebo; Drug: Itraconazole

INTERVENTIONS:
Drug: BAY1817080 — Study part 1: Escalating doses of BAY1817080; single dose administration; solid dosage form (redosing of BAY1817080 at dose group 1 and 2 together with itraconazole; redosing of BAY1817080 at dose group 4 together with food [American breakfast]) Study part 2: Escalating doses of BAY1817080; single dose administration together with an American breakfast; solid dosage form (redosing of BAY1817080 at dose group 1, 2 and 4 together with food [Continental breakfast])
  Arms: BAY1817080
Drug: Placebo — Study part 1: Escalating doses of respective placebos; single dose administration; solid dosage form (redosing of placebo at dose group 1 and 2 together with itraconazole; redosing of placebo at dose group 4 together with food [American breakfast]) Study part 2: Escalating doses of respective placebos; single dose administration together with an American breakfast; solid dosage form (redosing of placebo at dose group 1, 2 and together with food [Continental breakfast])
  Arms: Placebo
Drug: Itraconazole — Redosing of BAY1817080/placebo at dose group 1 and 2 together with itraconazole (study part 1)

SUMMARY:
This study is a first in human study that will investigate the safety, tolerability and pharmacokinetics of ascending single doses of BAY1817080 using a placebo controlled, randomized, single center design. In addition the influence of itraconazole and food on the pharmacokinetics of BAY1817080 will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* Age: 18 to 45 years (inclusive)
* Body mass index (BMI) : ≥18 and ≤30 kg/m²
* Race: White

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Relevant diseases within the last 4 weeks prior to the first drug administration
* Existing chronic diseases requiring medication
* Known or suspected malignant tumors or carcinoma in situ (including history of malignant tumors, with a status after treatment), known or suspected benign tumors of the liver and pituitary (including after treatment)
* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Use of any drugs which might influence the results of the trial within 14 days prior to administration or during the trial until follow-up including drugs which might affect the pharmacokinetics

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2017-05-11 (Actual); Study Completion 2017-08-23 (Actual)

PRIMARY OUTCOMES:
Frequency of treatment-emergent adverse events | Up to 4 months
Severity of treatment-emergent adverse events | Up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- CRS Clinical Research Services Berlin GmbH, Berlin, Germany

REFERENCES:
- [Derived] Reif S, Schultze-Mosgau MH, Engelen A, Piel I, Denner K, Roffel A, Tiessen R, Klein S, Francke K, Rottmann A. Mass Balance and Metabolic Pathways of Eliapixant, a P2X3 Receptor Antagonist, in Healthy Male Volunteers. Eur J Drug Metab Pharmacokinet. 2024 Jan;49(1):71-85. doi: 10.1007/s13318-023-00866-0. Epub 2023 Dec 3. PMID 38044419